CLINICAL TRIAL: NCT04001075
Title: A Phase I/IIa, Open-label, Dose-Escalation and Dose Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TJ107 in Chinese Patients With Advanced Solid Tumors
Brief Title: Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TJ107 in Chinese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ107001STM101
Record Dates: First submitted 2019-06-23; First posted 2019-06-27 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumord

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ107 (Experimental): Patients enrolled in dose escalation part will be given 2 doses (28 days/dose) during the main-treatment period
  Interventions: Drug: TJ107

INTERVENTIONS:
Drug: TJ107 — Patients enrolled in dose escalation part will be given 2 doses (28 days/dose) during the main-treatment period

SUMMARY:
This is a two-part study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of TJ107 in Chinese patients with advanced solid tumors. Approximately a total of 36 ~ 60 patients will be enrolled into the dose escalation cohorts (Part A), and expansion cohorts (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years old;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~2;
* Patients must have histological or cytological confirmation of advanced solid tumors that is refractory to standard therapy or for which there is no standard available therapy;
* Predicted life expectancy ≥3 months;
* Patients must have adequate organ and marrow function;
* Patients at reproductive age should take adequate contraceptive measures while on study drug and for 6 months following the last dose of study drug.
* Patients should have the ability and willingness to comply with the study and follow up. And patients must be able to provide written informed consent.

Exclusion Criteria:

* Patients who have experienced a Grade 3 or higher toxicity related to prior immunotherapy.
* Patients who are still receive anti-tumor therapy such as radiotherapy, chemotherapy, targeted therapy, endocrine therapy, or other clinical trials from 4 weeks prior to the first dose, or patients who have not recovered from previous toxicity to level 1.
* Women who are pregnant or breast feeding
* Patients who are drug-dependent or have a history of substance abuse or psychonosema history.
* Have been vaccinated within 4 weeks of study dosing, with the exception of licensed intranasal or intramuscular influenza vaccine during study
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Positive laboratory test for HBsAg with HBV DNA ≥ 100 IU/mL, or positive laboratory test for HCV.
* Prior treatment with immune checkpoint inhibitors, immunomodulatory mAbs, and/or mAb-derived therapies is allowed provided that at least 3 months or 5 half-lives of the drug, whichever is longer, have elapsed from the last dose.
* Uncontrolled concurrent illness.
* Major surgery procedure (excluding diagnostic surgery) within 4 weeks of the first dose of study drug.
* Patients with a history of treated CNS metastases.
* Other psychiatric illness/social situations that would limit compliance with the study requirements decided by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | 28days after first dose
  Safety and tolerability of TJ107. Incidence of dose-limiting toxicities (DLTs)
Adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Safety and tolerability of TJ107. Incidence of adverse events
Serious adverse events | through study completion, an average of 1 year
  Safety and tolerability of TJ107. Incidence of serious adverse events by National Cancer Institute Common Terminology Criteria for Adverse Events(CI CTCAE 5.0)

SECONDARY OUTCOMES:
Maximum tolerated dose | through study completion, an average of 1 year
  Maximum tolerated dose (MTD)
Maximum effective dose | through study completion, an average of 1 year
  Maximum effective dose (MED)
Recommended phase II dose | through study completion, an average of 1 year
  Recommended phase II dose (RP2D)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The sixth Affiliated Hospital, Sun Yat-sen University, Guanzhou, Guangdong
  - the First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, affiliated with the Zhejiang University School of the Medical, Hangzhou, Zhejiang